CLINICAL TRIAL: NCT03554135
Title: SAINT: Single frActIoN eighT Gray Palliative Radiotherapy With Modulated Intensity for Pain Reduction: a Single Arm Cohort Analysis
Brief Title: Single frActIoN eighT Gray Palliative Radiotherapy With Modulated Intensity for Pain Reduction
Acronym: SAINT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr. Cellini, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 0011201/18
Record Dates: First submitted 2018-05-31; First posted 2018-06-12 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Bone Metastases; Radiotherapy; Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Personalization of palliative radiotherapy — Observe the rates of pain control and the need to retreat patient, when applied to personalization of indications and maximum technological support for palliative radiotherapy to patients with < 6 months prognostic score attendance

SUMMARY:
Non-randomized, monocentric, observational study to evaluate the response in terms of reduction of painful symptoms from bone metastases to radiotherapy with high personalization of treatment: performed with modern technology, supplied with modulated intensity technique with concomitant integrated boost, according to selection of patients in accordance with prognosis determined by specific prognostic score

DETAILED DESCRIPTION:
Palliative antalgic oncological treatments concern a chronically-evolving disease patient with pain control problems, and are a complex problem from different points of view: logistic, clinical and scientific research. An increasing number of patients are afflicted due to the increased incidence of cancer in all its phases and the potential chronicity of the disease linked to new therapies.

The use of palliative anti-radiation radiotherapy treatments involves up to 40% of patients in a Radiotherapy Center. Radiotherapy was used in the palliative treatment of symptomatic bone metastases to improve quality of life (QoL) of these patients. This is the easiest way to respond to problems of home care or long-term care (eg: Hospice). This need is particularly accentuated for patients with a more severe situation. To reduce the overall duration of the treatment, it is necessary to manage hypofractionated regulators (ie with dose fractionation which daily dispense a dose higher than 2Gy). In fact, hypofractionated regimes concern the gold standard for these clinical presentations.

With the same pain control, multiple fractionation boards report better symptom control over time and are therefore very often preferred for patients with a prognosis> 6 months. On the other hand, the treatment regimen with 8 Gy in single therapy session is suggested as preferable for patients with a worse prognosis (ie less than 6 months of life expectancy). Evidence from literature suggests that palliative radiation therapy is effective in controlling pain even in the last weeks of the patient's life and therefore useful to improve the conditions of patients with a more severe prognosis.

The identification of patients with the worst prognosis to which single-agent radiotherapy is reserved is another crucial aspect. Unfortunately, although clinically validated in scientific trials, the routine use of prognostic scores is rarely used in everyday clinical practice to characterize life expectancy and define the most appropriate treatment regimen. This aspect limits the effective personalization of palliative treatments of this type.

Furthermore, the indications available in the literature do not specify a univocally shared standard of technical approach to radiant treatment. The Consensus Conference whose data have been reported by Chow et al. considers as potentially applicable both non-conformed techniques (e.g .: single back beam) and the most modern conformational techniques. The less conformed techniques have the defect of distributing in a more variable way the dose inside the target to irradiate and to save less well the organs at risk (OAR) with consequent increase of the risk of toxicity that could reduce the beneficial to the patient given by the reduction of pain from metastases.

Finally, the prescription of the single 8 Gy radiotherapy session in daily practice is still not sufficiently widespread, as evidenced by international literature . Due to the peculiar characteristics of the patients who need these treatments, scientific research aimed at optimizing these therapies is a need for assistance and even ethics.

This particular analysis, within the Umbrella Protocol, focuses on patients with uncomplicated and painful vertebral bone metastases, and is aimed at observing and recording the efficacy of treatment in a single 8 Gy session, applied in good clinical practice. according to available evidence.

Particular attention is paid to applying a high degree of personalization of the treatment and a modern approach to the technology of performing the radiant treatment. The personalization of the treatment will be favored by the routine use of: i) a valid prognostic score for the expected survival, the Mizumoto prognostic Score (Mizumoto M, 2008), to identify patients with the worst prognosis to offer treatment in a single session. The use of the most advanced radiation dose administration technologies will be applied by choosing (in the spectrum of technologies applicable to these clinical presentations) the most modern modulated intensity radiotherapy (IMRT). IMRT allows to reduce the dose administered to the OAR and to concentrate the areas with the highest dose concentration (the so-called "hot spots") only within the evidence of disease (or "Gross tumor Volume" - GTV). Through the integrated simultaneous boost (SIB) method in IMRT, it is possible, in fact, to check the extent and location of the "hot zones" by specifying, through precise prescription, the maximum desired amount and the topographic limits to the inside of the target prescribed at the dose of 8 Gy, however doing "drop" the dose to the surrounding OAR.

The hypothesis of the study is to observe the rates of pain control and the need to retract the patient, when applied to personalization of indications and maximum technological support. These results could be a basis of scientific evidence to further support the clinical orientation towards the use of the single fraction of radiotherapy with consequent improvement in the quality of life of these patients. Furthermore, such data will be able to feed further analyzes aimed at the cost / effectiveness of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with spinal bone metastases from solid, uncomplicated tumor
* Established primary or secondary tumor histology correlated to the treatment lesion
* Age >18 years
* Obtaining informed consent
* Symptomatic patients (NRS> = 4) at the treatment site
* Prognosis <6 months according to Mizumoto Prognostic Score (i.e. Class B or C)
* Spine Instability Neoplastic Score (SINS) <7

Exclusion Criteria:

* Concurrent disorders (psychiatric and otherwise) which, in the opinion of the investigator, make data collection unreliable
* Impossibility to assign specific NRS for each CTV to be enrolled
* Previous radiotherapy at the same site or at the level of adjoining metamers (higher or lower than the one to be enrolled)
* Radiometabolic therapy
* Previous enrollment of the same patient for 3 irradiated lesions
* Epidural compression of the spinal cord or of the cauda equina
* Injuries affecting> 25% of the medullary canal and / or a distance <5 mm from the medulla or from the cauda
* Injuries with indication of surgical stabilization
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Considering the observational nature of the study, all patients corresponding to the "Inclusion Criteria" will be taken into consideration over a period of 6 months from the beginning of the study. 50 patients are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain control | 1 month after end of radiotherapy
  Pain control measured with Numeric Rating Scale (NRS) score, a 11-point scale for patient self-reporting of pain.
  NRS score presents a total range between 0 (no pain) and 10 maximum pain.
  NRS subscale are the sequent:
  * 0: no pain
  * 1-3: mild pain
  * 4-6: moderate pain
  * 7-10 severe pain

SECONDARY OUTCOMES:
Re-treatment during follow up | 12 months after end of radiotherapy
  Rate of re-treatment during follow up
Pain-dipendent variables | 12 months after end of radiotherapy
  To evaluate the possible correlation between the adequacy of antalgic treatment and potential predictors such as tumor type, purpose of treatment, care setting, stage of disease

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cellini, MD, Principal Investigator — Fondazione Policlinico Gemelli IRCCS - Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Result] Bentzen SM, Constine LS, Deasy JO, Eisbruch A, Jackson A, Marks LB, Ten Haken RK, Yorke ED. Quantitative Analyses of Normal Tissue Effects in the Clinic (QUANTEC): an introduction to the scientific issues. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S3-9. doi: 10.1016/j.ijrobp.2009.09.040. PMID 20171515
- [Result] Braam P, Lambin P, Bussink J. Stereotactic versus conventional radiotherapy for pain reduction and quality of life in spinal metastases: study protocol for a randomized controlled trial. Trials. 2016 Feb 2;17:61. doi: 10.1186/s13063-016-1178-7. PMID 26829933
- [Result] Chow E, Hoskin P, Mitera G, Zeng L, Lutz S, Roos D, Hahn C, van der Linden Y, Hartsell W, Kumar E; International Bone Metastases Consensus Working Party. Update of the international consensus on palliative radiotherapy endpoints for future clinical trials in bone metastases. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1730-7. doi: 10.1016/j.ijrobp.2011.02.008. Epub 2011 Apr 12. PMID 21489705
- [Result] Correa RJ, Salama JK, Milano MT, Palma DA. Stereotactic Body Radiotherapy for Oligometastasis: Opportunities for Biology to Guide Clinical Management. Cancer J. 2016 Jul-Aug;22(4):247-56. doi: 10.1097/PPO.0000000000000202. PMID 27441744
- [Result] Deodato F, Cilla S, Macchia G, Torre G, Caravatta L, Mariano G, Mignogna S, Ferro M, Mattiucci GC, Balducci M, Frascino V, Piermattei A, Ferrandina G, Valentini V, Morganti AG. Stereotactic radiosurgery (SRS) with volumetric modulated arc therapy (VMAT): interim results of a multi-arm phase I trial (DESTROY-2). Clin Oncol (R Coll Radiol). 2014 Dec;26(12):748-56. doi: 10.1016/j.clon.2014.08.005. Epub 2014 Aug 29. PMID 25175042
- [Result] Furfari A, Wan BA, Ding K, Wong A, Zhu L, Bezjak A, Wong R, Wilson CF, DeAngelis C, Azad A, Chow E, Charames GS. Genetic biomarkers associated with pain flare and dexamethasone response following palliative radiotherapy in patients with painful bone metastases. Ann Palliat Med. 2017 Dec;6(Suppl 2):S240-S247. doi: 10.21037/apm.2017.09.04. Epub 2017 Sep 20. PMID 29156912
- [Result] Guckenberger M, Hawkins M, Flentje M, Sweeney RA. Fractionated radiosurgery for painful spinal metastases: DOSIS - a phase II trial. BMC Cancer. 2012 Nov 19;12:530. doi: 10.1186/1471-2407-12-530. PMID 23164174
- [Result] Mizumoto M, Harada H, Asakura H, Hashimoto T, Furutani K, Hashii H, Takagi T, Katagiri H, Takahashi M, Nishimura T. Prognostic factors and a scoring system for survival after radiotherapy for metastases to the spinal column: a review of 544 patients at Shizuoka Cancer Center Hospital. Cancer. 2008 Nov 15;113(10):2816-22. doi: 10.1002/cncr.23888. PMID 18846565
- [Result] Murai T, Murata R, Manabe Y, Sugie C, Tamura T, Ito H, Miyoshi Y, Shibamoto Y. Intensity modulated stereotactic body radiation therapy for single or multiple vertebral metastases with spinal cord compression. Pract Radiat Oncol. 2014 Nov-Dec;4(6):e231-7. doi: 10.1016/j.prro.2014.02.005. Epub 2014 Mar 31. PMID 25407874
- [Result] Ryu S, Pugh SL, Gerszten PC, Yin FF, Timmerman RD, Hitchcock YJ, Movsas B, Kanner AA, Berk LB, Followill DS, Kachnic LA. RTOG 0631 phase 2/3 study of image guided stereotactic radiosurgery for localized (1-3) spine metastases: phase 2 results. Pract Radiat Oncol. 2014 Mar-Apr;4(2):76-81. doi: 10.1016/j.prro.2013.05.001. Epub 2013 Jun 4. PMID 24890347
- [Result] van der Velden JM, Verkooijen HM, Seravalli E, Hes J, Gerlich AS, Kasperts N, Eppinga WS, Verlaan JJ, van Vulpen M. Comparing conVEntional RadioTherapy with stereotactIC body radiotherapy in patients with spinAL metastases: study protocol for an randomized controlled trial following the cohort multiple randomized controlled trial design. BMC Cancer. 2016 Nov 21;16(1):909. doi: 10.1186/s12885-016-2947-0. PMID 27871280